CLINICAL TRIAL: NCT05849142
Title: Feasibility of Adaptive Radiation Therapy for Human-papilloma Virus-positive Oropharyngeal Cancer Patients on MRIdian Linac
Acronym: OPC-V
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: MRI Linac contract was not renewed at our institution after Viewray went bankrupt. Therefore we cannot do adaptive treatments on this machine. No patients were enrolled.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Stuart Samuels, Associate Professor of Clinical Medicine, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220776
Record Dates: First submitted 2023-04-25; First posted 2023-05-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Oropharynx Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MRIdian Linac Group (Experimental): All accrued participants will be enrolled onto the MRIdian Linac Group. Participants will receive adaptive radiotherapy (ART) on the MRIdian Linac. Participants will complete the duration of their radiotherapy regimen on the MRIdian Linac for approximately 7 weeks.
  Interventions: Device: MRIdian Linac

INTERVENTIONS:
Device: MRIdian Linac — Radiation therapy (RT) will be delivered with an integrated MRI-RT delivery system (MRIdian Linac). Participants will then receive standard-of-care RT with a dose prescription of 70 Gy in 35 fractions on the MRIdian Linac. Adaptive RT (ART) planning will occur every 5th fraction of RT.
  Other Names: ViewRay

SUMMARY:
The purpose of this research is to determine whether it is feasible to treat patients with Human Papilloma Virus positive (HPV-positive) oropharyngeal tumors on a specialized treatment machine (MRIdian linear accelerator [Linac]), which utilizes magnetic resonance imaging (MRI) for radiation planning and delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed new diagnosis of HPV-positive OPC [i.e. Base of tongue, tonsil, soft palate, vallecula, and posterior pharyngeal wall]
* American Joint Committee on Cancer (AJCC) 8th edition Stage I-III planned for definitive chemoradiation.
* Members of all races and ethnic backgrounds
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for duration of study participation.
* Must be able to understand and sign an Institutional Review Board (IRB)-approved written informed consent document.

Exclusion Criteria:

* Prior surgery, chemotherapy, or radiation treatment for head and neck cancer
* Prior history of cancer other than non-melanomatous skin cancer
* Distant metastases (cM1) or (pM1) disease)
* Evidence of a compromised airway
* Medical contraindications to MRIs
* Unable to tolerate MRIs without sedation
* Pregnant patients
* Breastfeeding patients
* Eastern Cooperative Oncology Group (ECOG) performance status >1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent difference between initial reference plan and adaptive weekly RT plan | Up to 6 months
  Weekly adaptive plans will be compared to the initial reference plan and compared using a percent difference equation estimating the actual values of the quantities used as dosimetric constraints for each participant between the initial reference plan and the weekly adaptive plan[s].
Evaluation of deformable imaging registration | Up to 6 months
  For evaluation of deformable imaging registration, deformed contours will be compared to the physician-segmented contours using the Dice similarity coefficient (DSC).

SECONDARY OUTCOMES:
Treatment times recorded in minutes | Up to 6 months
  We will follow previously-established guidelines by the MR-Linac Consortium Head and Neck Tumor Site for measuring treatment times. Treatment times will be calculated in minutes from the time stamps in the record and verify system. Three timepoints will be recorded: [1] setup and plan optimization [i.e. time between the participant's arrival to the MRidian and delivery of the first beam]; [2] beam delivery [i.e. the time between delivery of the first and last beam]; and [3] total treatment time.
Patient-reported Quality of Life as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ) (EORTC QLQ-C30) | Up to 1 year
  Quality of life will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). It consists of 30 items to measure multiple aspects that incorporated five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea/vomiting), a global health status/QoL scale, and six single common items (dyspnea, loss of appetite, insomnia, constipation, diarrhea, and financial difficulties). The scoring system ranged from 1 (not at all) to 4 (very much). High scores for functional items and low scores for symptoms represent the good QoL.There are two questions for the overall quality of life rating, and the ranking ranged from 1 (very poor) to 7 (excellent).
Patient-reported Quality of Life as measured by the European Organization for Research and Treatment Head & Neck 43 | Up to 1 year
  Quality of life will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-H&N43). The questionnaire used will be for that for head and neck patients, score range from 1 (not at all) to 4 (very much), higher scores indicate lower quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Samuels, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- The University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No